CLINICAL TRIAL: NCT05342753
Title: A Prospective Clinical Study to Evaluate Safety and Effectiveness of Restylane® Kysse for Lip Augmentation in Chinese Subjects
Brief Title: Safety and Effectiveness of Restylane® Kysse for Lip Augmentation in Chinese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05DF2007
Record Dates: First submitted 2022-03-16; First posted 2022-04-25 (Actual); Results first posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Lip Augmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Restylane Kysse (Experimental): Hyaluronic Acid
  Interventions: Device: Restylane Kysse

INTERVENTIONS:
Device: Restylane Kysse — Hyaluronic Acid: Injectable gel for lip augmentation and the correction of upper perioral rhytids

SUMMARY:
Open-label, phase IV, post-marketing study to evaluate aesthetic improvement in Chinese subjects after treatment with Restylane Kysse.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing to comply with the requirements of the study and providing a signed written informed consent
* Ability to adequately understand the verbal explanations and the written subject information provided in English
* Subjects seeking augmentation therapy for the lips
* Adult males or non-pregnant, non-breastfeeding females, 22 years of age or older with both biological parents of full Chinese descent

Exclusion Criteria:

* Known/previous allergy or hypersensitivity to any injectable hyaluronic acid (HA) gel or to gram-positive bacterial proteins
* Previous use of any permanent (non-biodegradable) or semipermanent (e.g., calcium hydroxylapatite or poly-L-lactic acid) facial tissue augmentation therapy, lifting threads, permanent implants or autologous fat below the level of the lower orbital rim.
* Previous use of any HA-based or collagen-based biodegradable facial tissue augmentation therapy below the level of the lower orbital rim within 12 months prior to the baseline visit.
* Previous facial surgery, within 6 months, below the level of the lower orbital rim
* Previous surgery to the upper or lower lip, lip piercing or tattoo, or history of facial trauma.
* Participation in any interventional clinical study within 30 days of screening

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Galderma R&D
Locations (3):
- United States (3):
  - Galderma Research Site, Los Angeles, California
  - Galderma Research Site, Vista, California
  - Galderma Research Site, Ardmore, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 13 June 2022 to 07 November 2024.
Pre-assignment Details: A total of 25 participants with a score of 1 (Very Thin) or 2 (Thin) on the Medicis Lip Fullness Scale (MLFS) were screened for the study, of which 3 were screen failures. 22 participants were treated with Restylane Kysse in at least 1 lip.
Groups:
- Restylane Kysse: Participants received an injection in the lips with sufficient amount of Restylane Kysse to achieve optimal aesthetic improvement, as determined by the Investigator and participant at baseline (Day 1) with optional touch-up treatments at the 4-week follow-up visit.
Period: Overall Study
Arm/Group | Restylane Kysse
Started | 22
Completed | 15
Not Completed | 7
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who were treated with Restylane Kysse in at least 1 lip and were analyzed according to the treatment actually received.
Arm/Group | Restylane Kysse
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 22
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han Chinese | 22
MLFS-upper lip [Count of Participants; unit: Participants]
  1 (very thin) | 0
  2 (thin) | 22
MLFS-lower lip [Count of Participants; unit: Participants]
  1 (very thin) | 0
  2 (thin) | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Assessed as At Least 1-point Improvement From Baseline on Medicis Lip Fullness Scale (MLFS)
Description: The MLFS is a validated photograph-based outcome instrument that is designed specifically for quantifying lip fullness. Scoring of lip fullness from Grade 1 to 5 (grade 1: "Very Thin", grade 2: "Thin", grade 3: "Medium", grade 4: "Full" and grade 5: "Very Full"; with a higher score reflecting greater lip fullness) was based on visual live assessment by the Investigator. Percentage of participants with at least 1-point improvement from baseline on MLFS are reported for this outcome measure.
Time Frame: At Week 8
Population: The modified intent-to-treat (mITT) population included all participants who were treated in both lips. Here, 'overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Restylane Kysse
Number analyzed (Participants) | 19
percentage of participants
  Upper lip | 94.7
  Lower lip | 94.7

2. Primary Outcome: Percentage of Participants Assessed as At Least 1-point Improvement From Baseline on MLFS
Description: as for outcome 1
Time Frame: At Week 16
Population: The mITT population included all participants who were treated in both lips. Here, 'overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Restylane Kysse
Number analyzed (Participants) | 17
percentage of participants
  Upper lip | 94.1
  Lower lip | 94.1

3. Primary Outcome: Percentage of Participants Assessed as At Least 1-point Improvement From Baseline on MLFS
Description: as for outcome 1
Time Frame: At Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Restylane Kysse
Number analyzed (Participants) | 14
percentage of participants
  Upper lip | 92.9
  Lower lip | 92.9

4. Primary Outcome: Percentage of Participants Assessed as At Least 1-point Improvement From Baseline on MLFS
Description: as for outcome 1
Time Frame: At Week 32
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Restylane Kysse
Number analyzed (Participants) | 16
percentage of participants
  Upper lip | 87.5
  Lower lip | 87.5

5. Primary Outcome: Percentage of Participants Assessed as At Least 1-point Improvement From Baseline on MLFS
Description: as for outcome 1
Time Frame: At Week 40
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Restylane Kysse
Number analyzed (Participants) | 15
percentage of participants
  Upper lip | 86.7
  Lower lip | 86.7

6. Primary Outcome: Percentage of Participants Assessed as At Least 1-point Improvement From Baseline on MLFS
Description: as for outcome 1
Time Frame: At Week 48
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Restylane Kysse
Number analyzed (Participants) | 15
percentage of participants
  Upper lip | 86.7
  Lower lip | 86.7

7. Primary Outcome: Change From Baseline on the MLFS by Treatment Area at Week 8 After the Last Injection
Description: The MLFS is a validated photograph-based outcome instrument that is designed specifically for quantifying lip fullness. Scoring of lip fullness from Grade 1 to 5 (grade 1: "Very Thin", grade 2: "Thin", grade 3: "Medium", grade 4: "Full" and grade 5: "Very Full"; with a higher score reflecting greater lip fullness) was based on visual live assessment by the Investigator. Improvement was defined as at least 1-point change from baseline in lip fullness. Number of participants with no improvement, one grade, two grade and three grade improvement are reported for this outcome measure.
Time Frame: 8 weeks after last injection (up to 12 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Kysse
Number analyzed (Participants) | 19
Participants
  Upper lip: No improvement | 1
  Upper lip: One grade improvement | 10
  Upper lip: Two grade improvement | 7
  Upper lip: Three grade improvement | 1
  Lower lip: No improvement | 1
  Lower lip: One grade improvement | 8
  Lower lip: Two grade improvement | 9
  Lower lip: Three grade improvement | 1

8. Primary Outcome: Change From Baseline on the MLFS by Treatment Area at Week 16 After the Last Injection
Description: as for outcome 7
Time Frame: 16 weeks after last injection (up to 20 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Kysse
Number analyzed (Participants) | 17
Participants
  Upper lip: No improvement | 1
  Upper lip: One grade improvement | 7
  Upper lip: Two grade improvement | 8
  Upper lip: Three grade improvement | 1
  Lower lip: No improvement | 1
  Lower lip: One grade improvement | 6
  Lower lip: Two grade improvement | 9
  Lower lip: Three grade improvement | 1

9. Primary Outcome: Change From Baseline on the MLFS by Treatment Area at Week 24 After the Last Injection
Description: as for outcome 7
Time Frame: 24 weeks after last injection (up to 28 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Kysse
Number analyzed (Participants) | 14
Participants
  Upper lip: No improvement | 1
  Upper lip: One grade improvement | 6
  Upper lip: Two grade improvement | 6
  Upper lip: Three grade improvement | 1
  Lower lip: No improvement | 1
  Lower lip: One grade improvement | 6
  Lower lip: Two grade improvement | 6
  Lower lip: Three grade improvement | 1

10. Primary Outcome: Change From Baseline on the MLFS by Treatment Area at Week 32 After the Last Injection
Description: as for outcome 7
Time Frame: 32 weeks after last injection (up to 36 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Kysse
Number analyzed (Participants) | 16
Participants
  Upper lip: No improvement | 2
  Upper lip: One grade improvement | 9
  Upper lip: Two grade improvement | 4
  Upper lip: Three grade improvement | 1
  Lower lip: No improvement | 2
  Lower lip: One grade improvement | 8
  Lower lip: Two grade improvement | 5
  Lower lip: Three grade improvement | 1

11. Primary Outcome: Change From Baseline on the MLFS by Treatment Area at Week 40 After the Last Injection
Description: as for outcome 7
Time Frame: 40 weeks after last injection (up to 44 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Kysse
Number analyzed (Participants) | 15
Participants
  Upper lip: No improvement | 2
  Upper lip: One grade improvement | 8
  Upper lip: Two grade improvement | 4
  Upper lip: Three grade improvement | 1
  Lower lip: No improvement | 2
  Lower lip: One grade improvement | 7
  Lower lip: Two grade improvement | 5
  Lower lip: Three grade improvement | 1

12. Primary Outcome: Change From Baseline on the MLFS by Treatment Area at Week 48 After the Last Injection
Description: as for outcome 7
Time Frame: 48 weeks after last injection (up to 52 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Kysse
Number analyzed (Participants) | 15
Participants
  Upper lip: No improvement | 2
  Upper lip: One grade improvement | 9
  Upper lip: Two grade improvement | 4
  Upper lip: Three grade improvement | 0
  Lower lip: No improvement | 2
  Lower lip: One grade improvement | 9
  Lower lip: Two grade improvement | 4
  Lower lip: Three grade improvement | 0

13. Secondary Outcome: Percentage of Responders With At Least "Improved" on the Wrinkle Assessment Scale (WAS)
Description: The WAS is a validated photograph-based outcome instrument that is designed specifically for quantifying facial folds. Scoring of fold severity is based on visual assessment of the length and apparent depth of the wrinkle at a certain time-point. Scoring of the upper perioral rhytids and oral commissures was based on visual live assessment by the investigator at defined time points; by using respective categorical scale ranging from Grade 0 to 5 where: grade 0 or 'No wrinkles', (1) 'Just perceptible wrinkle', (2) 'Shallow wrinkles', (3) 'Moderately deep wrinkle', (4) 'Deep wrinkle, well-defined edges', (5) 'Very deep wrinkle, redundant fold', higher grade represented higher fold severity. Responder was defined as a participant with at least a 1-point improvement from baseline.
Time Frame: At Weeks 8, 16, 24, 32, 40, and 48
Population: The mITT population included all participants who were treated in both lips. Here, 'number analyzed' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Restylane Kysse
Number analyzed (Participants) | 22
percentage of participants
  Upper perioral rhytids; Week 8: number analyzed (Participants) | 2
  Upper perioral rhytids; Week 8 | 100 [15.8 to 100.0]
  Upper perioral rhytids; Week 16: number analyzed (Participants) | 1
  Upper perioral rhytids; Week 16 | 100 [2.5 to 100.0]
  Upper perioral rhytids; Week 24: number analyzed (Participants) | 1
  Upper perioral rhytids; Week 24 | 100.0 [2.5 to 100.0]
  Upper perioral rhytids; Week 32: number analyzed (Participants) | 1
  Upper perioral rhytids; Week 32 | 100.0 [2.5 to 100.0]
  Upper perioral rhytids; Week 40: number analyzed (Participants) | 1
  Upper perioral rhytids; Week 40 | 100.0 [2.5 to 100.0]
  Upper perioral rhytids; Week 48: number analyzed (Participants) | 1
  Upper perioral rhytids; Week 48 | 100.0 [2.5 to 100.0]
  Left oral commissures; Week 8: number analyzed (Participants) | 13
  Left oral commissures; Week 8 | 92.3 [64.0 to 99.8]
  Left oral commissures; Week 16: number analyzed (Participants) | 12
  Left oral commissures; Week 16 | 100.0 [73.5 to 100.0]
  Left oral commissures; Week 24: number analyzed (Participants) | 11
  Left oral commissures; Week 24 | 90.9 [58.7 to 99.8]
  Left oral commissures; Week 32: number analyzed (Participants) | 12
  Left oral commissures; Week 32 | 91.7 [61.5 to 99.8]
  Left oral commissures; Week 40: number analyzed (Participants) | 11
  Left oral commissures; Week 40 | 100.0 [71.5 to 100.0]
  Left oral commissures; Week 48: number analyzed (Participants) | 11
  Left oral commissures; Week 48 | 100.0 [71.5 to 100.0]
  Right oral commissures; Week 8: number analyzed (Participants) | 13
  Right oral commissures; Week 8 | 92.3 [64.0 to 99.8]
  Right oral commissures; Week 16: number analyzed (Participants) | 12
  Right oral commissures; Week 16 | 100.0 [73.5 to 100.0]
  Right oral commissures; Week 24: number analyzed (Participants) | 11
  Right oral commissures; Week 24 | 90.9 [58.7 to 99.8]
  Right oral commissures; Week 32: number analyzed (Participants) | 12
  Right oral commissures; Week 32 | 91.7 [61.5 to 99.8]
  Right oral commissures; Week 40: number analyzed (Participants) | 11
  Right oral commissures; Week 40 | 100.0 [71.5 to 100.0]
  Right oral commissures; Week 48: number analyzed (Participants) | 11
  Right oral commissures; Week 48 | 100.0 [71.5 to 100.0]

14. Secondary Outcome: Percentage of Participants With At Least "Improved" on the Global Aesthetic Improvement Scale (GAIS) as Assessed by Treating Investigator at Weeks 8, 16, 24, 32, 40, and 48
Description: The GAIS is a 7-point categorical scale ranging from -3 (Very Much Worse) to +3 (very much improved), used by the Treating Investigator to assess changes in the appearance of participants' lips following treatment by responding to the question: "With respect to the appearance of the participant's lips, how would you describe the result of the lip treatment compared to the photos taken before treatment?" by using the respective categorical scale as follows: Very Much Improved, Much Improved, Improved, No Change, Worse, Much Worse, Very Much Worse. In this outcome measure, percentage of participants who achieved at least 'Improved' on the GAIS assessed by treating investigator at Weeks 8, 16, 24, 32, 40, and 48 were reported.
Time Frame: At Weeks 8, 16, 24, 32, 40, and 48
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Restylane Kysse
Number analyzed (Participants) | 22
percentage of participants
  At Week 8: number analyzed (Participants) | 19
  At Week 8 | 100.0 [82.4 to 100.0]
  At Week 16: number analyzed (Participants) | 17
  At Week 16 | 100.0 [80.5 to 100.0]
  At Week 24: number analyzed (Participants) | 14
  At Week 24 | 100.0 [76.8 to 100.0]
  At Week 32: number analyzed (Participants) | 16
  At Week 32 | 100.0 [79.4 to 100.0]
  At Week 40: number analyzed (Participants) | 15
  At Week 40 | 100.0 [78.2 to 100.0]
  At Week 48: number analyzed (Participants) | 15
  At Week 48 | 100.0 [78.2 to 100.0]

ADVERSE EVENTS:
Time Frame: From Visit 1 of the study up to follow-up visit (Week 48)
Description: The safety population included all subjects who were treated with Restylane Kysse in at least 1 lip and were analyzed according to the treatment actually received.
Arm/Group | Restylane Kysse
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 2/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Restylane Kysse (N=22)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT05342753/Prot_002.pdf
  • Statistical Analysis Plan (2023-10-06): https://cdn.clinicaltrials.gov/large-docs/53/NCT05342753/SAP_003.pdf